CLINICAL TRIAL: NCT00910819
Title: Prospective and Retrospective Observation of the Adjuvant and Palliative Treatment Strategies in the Therapy of Colorectal Cancer in Germany
Brief Title: Tumour Registry Colorectal Cancer
Acronym: TKK
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: Arbeitskreis Klinische Studien (Other); Arbeitsgemeinschaft fur Internistische Onkologie (Other)
Responsible Party: Sponsor
Other Study IDs: IOM TKK
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Advanced Colorectal Cancer; Epidemiology; Health Services Research; Germany; Registry; Palliative Care; Palliative Treatment; Adjuvant Drug Therapy; Nutrition Assessment; Physical Activity
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
To describe treatment reality of patients with colorectal cancer treated by office-based and clinic-based medical oncologists in Germany.

DETAILED DESCRIPTION:
The TKK is a prospective, longitudinal, nation wide cohort study with the purpose to record information on the antineoplastic treatment of colorectal cancer in Germany. The registry will follow patients for up to five years. It will identify common therapeutic sequences and changes in the treatment of the disease. At inclusion, data in patient characteristics, comorbidities, tumor characteristics, biomarker testing and previous treatments are collected. During the course of observation data on all systemic treatments, radiotherapies, surgeries, and outcome are documented.

The impact of nutrition (CoNut) and physical activity (CoNut) on the course of the adjuvant disease will be examined, as well as long-term effects of adjuvant treatment (CoTox) and the final phase of the palliative process (CoLife). Based on the available data a prognostic score will be developed.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer
* 18 years and older
* Antineoplastic treatment

Exclusion Criteria:

* No colorectal cancer
* Below 18 years
* No antineoplastic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients undergoing antineoplastic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Course of Antineoplastic Treatment | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Roland Schnell, MD, Study Chair
Locations (1):
- iOMEDICO AG, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marschner N, Arnold D, Engel E, Hutzschenreuter U, Rauh J, Freier W, Hartmann H, Frank M, Janicke M. Oxaliplatin-based first-line chemotherapy is associated with improved overall survival compared to first-line treatment with irinotecan-based chemotherapy in patients with metastatic colorectal cancer - Results from a prospective cohort study. Clin Epidemiol. 2015 Apr 20;7:295-303. doi: 10.2147/CLEP.S73857. eCollection 2015. PMID 25945067
- [Background] Marschner N, Frank M, Vach W, Ladda E, Karcher A, Winter S, Janicke M, Trarbach T. Development and validation of a novel prognostic score to predict survival in patients with metastatic colorectal cancer: the metastatic colorectal cancer score (mCCS). Colorectal Dis. 2019 Jul;21(7):816-826. doi: 10.1111/codi.14600. Epub 2019 Mar 18. PMID 30834622